CLINICAL TRIAL: NCT02893501
Title: An Exploratory Study to Evaluate the Microbial Consortia of Infants (9-12 Months) Experiencing Diaper Rash and When Healthy
Brief Title: Infant Microbiome in Diaper Rash
Status: Completed | Type: Observational
Sponsor: Kimberly-Clark Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 500-16-0002
Record Dates: First submitted 2016-08-29; First posted 2016-09-08 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Diaper Rash
MeSH Terms: conditions — Diaper Rash

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: None Retained — swabs and tape strips of the diaper rash area will be analyzed
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to evaluate the microbiome composition of infant's (9-12 month) skin experiencing diaper rash in order to determine if the onset and severity of erythema associated with diaper rash is influenced by the type of bacteria colonizing the skin.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 9-12 months with mild to moderate diaper rash

Exclusion Criteria:

* Use of topical or oral antibiotics or antifungals within the past 4 weeks.
* Use of zinc-containing diaper rash creams within 48 hours first sample
* Immunocompromised

Ages: 9 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Community sample of male and female infants with mild to moderate diaper rash
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-09; Primary Completion 2017-01-04 (Actual); Study Completion 2017-01-04 (Actual)

PRIMARY OUTCOMES:
Operational Taxonomic Units (OTUs) of microbes present on skin | Change from Baseline at Day 14
Relative abundance of microbes present on skin measured in picograms of DNA | Change from Baseline at Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Sahra Niazi, MD, Principal Investigator — Midwest Children's Health Research Institute
Locations (1):
- Midwest Children's Health Research Institute, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costello EK, Lauber CL, Hamady M, Fierer N, Gordon JI, Knight R. Bacterial community variation in human body habitats across space and time. Science. 2009 Dec 18;326(5960):1694-7. doi: 10.1126/science.1177486. Epub 2009 Nov 5. PMID 19892944
- [Background] Le Lamer M, Pellerin L, Reynier M, Cau L, Pendaries V, Leprince C, Mechin MC, Serre G, Paul C, Simon M. Defects of corneocyte structural proteins and epidermal barrier in atopic dermatitis. Biol Chem. 2015 Nov;396(11):1163-79. doi: 10.1515/hsz-2015-0141. PMID 26020560
- [Background] Sakabe J, Kamiya K, Yamaguchi H, Ikeya S, Suzuki T, Aoshima M, Tatsuno K, Fujiyama T, Suzuki M, Yatagai T, Ito T, Ojima T, Tokura Y. Proteome analysis of stratum corneum from atopic dermatitis patients by hybrid quadrupole-orbitrap mass spectrometer. J Allergy Clin Immunol. 2014 Oct;134(4):957-60.e8. doi: 10.1016/j.jaci.2014.07.054. No abstract available. PMID 25282569
- [Background] Adalat S, Wall D, Goodyear H. Diaper dermatitis-frequency and contributory factors in hospital attending children. Pediatr Dermatol. 2007 Sep-Oct;24(5):483-8. doi: 10.1111/j.1525-1470.2007.00499.x. PMID 17958792